CLINICAL TRIAL: NCT02618967
Title: A Randomized, Double Blind Placebo Controlled, First in Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Subcutaneous Doses of AMG 570 in Healthy Subjects
Brief Title: Single Ascending Dose Study of AMG 570 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20140322
Record Dates: First submitted 2015-10-13; First posted 2015-12-02 (Estimated); Results first posted 2021-10-15 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Healthy Volunteer; Safety Study; Placebo Control; Phase 1
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — rozibafusp alfa; Drug Evaluation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- AMG 570 - 7 mg (Experimental): Participants will receive a single dose 7 mg dose of AMG 570 administered subcutaneously.
  Interventions: Biological: AMG 570
- AMG 570 - 21 mg (Experimental): Participants will receive a single 21 mg dose of AMG 570 administered subcutaneously.
  Interventions: Biological: AMG 570
- AMG 570 - 70 mg (Experimental): Participants will receive a single 70 mg dose of AMG 570 administered subcutaneously.
  Interventions: Biological: AMG 570
- AMG 570 - 140 mg (Experimental): Participants will receive a single 140 mg dose of AMG 570 administered subcutaneously.
  Interventions: Biological: AMG 570
- AMG 570 - 210 mg (Experimental): Participants will receive a single 210 mg dose of AMG 570 administered subcutaneously.
  Interventions: Biological: AMG 570
- AMG 570 - 420 mg (Experimental): Participants will receive a single 420 mg dose of AMG 570 administered subcutaneously.
  Interventions: Biological: AMG 570
- AMG 570 - 700 mg (Experimental): Participants will receive a single 700 mg dose of AMG 570 administered subcutaneously.
  Interventions: Biological: AMG 570
- Placebo (Placebo Comparator): Participants will receive a single dose of the matching AMG 570 placebo administered subcutaneously.
  Interventions: Biological: AMG 570 Matching Placebo

INTERVENTIONS:
Biological: AMG 570 — 7 dose levels of AMG 570 administered as single dose subcutaneous in healthy volunteers.
  Other Names: Active Comparator, Investigational Product, and Study drug
  Arms: AMG 570 - 140 mg; AMG 570 - 21 mg; AMG 570 - 210 mg; AMG 570 - 420 mg; AMG 570 - 7 mg; AMG 570 - 70 mg; AMG 570 - 700 mg
Biological: AMG 570 Matching Placebo — Placebo administered as single dose subcutaneous in healthy volunteers.
  Other Names: Placebo, Investigational Product, and Study drug
  Arms: Placebo

SUMMARY:
The purpose of this study is to obtain initial information on the safety and tolerability (effects good or bad), pharmacokinetics (what the body does to the drug), and pharmacodynamics (what the drug does to the body) of a single dose of AMG 570.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the investigator
* Normal or clinically acceptable electrocardiogram (ECG)
* Female subjects must be of documented non-reproductive potential
* Subjects must be current for all vaccinations
* Other inclusion criteria may apply

Exclusion Criteria:

* Current or chronic history of liver disease
* History of active infections
* History of significant respiratory disorder
* Evidence of renal disease
* Other exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Research Site, Evansville, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Abuqayyas L, Chen PW, Dos Santos MT, Parnes JR, Doshi S, Dutta S, Houk BE. Pharmacokinetics and Pharmacokinetic/Pharmacodynamic Properties of Rozibafusp Alfa, a Bispecific Inhibitor of BAFF and ICOSL: Analyses of Phase I Clinical Trials. Clin Pharmacol Ther. 2023 Aug;114(2):371-380. doi: 10.1002/cpt.2929. Epub 2023 May 24. PMID 37150935
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 56 healthy participants were enrolled at 3 research centers in the United States from 28 March 2016 to 06 September 2018.
Groups:
- AMG 570 - 7 mg: Participants received a single dose 7 mg dose of AMG 570 administered subcutaneously.
- AMG 570 - 21 mg: Participants received a single 21 mg dose of AMG 570 administered subcutaneously.
- AMG 570 - 70 mg: Participants received a single 70 mg dose of AMG 570 administered subcutaneously.
- AMG 570 - 140 mg: Participants received a single 140 mg dose of AMG 570 administered subcutaneously.
- AMG 570 - 210 mg: Participants received a single 210 mg dose of AMG 570 administered subcutaneously.
- AMG 570 - 420 mg: Participants received a single 420 mg dose of AMG 570 administered subcutaneously.
- AMG 570 - 700 mg: Participants received a single 700 mg dose of AMG 570 administered subcutaneously.
- Placebo: Participants received a single dose of the matching AMG 570 placebo administered subcutaneously.
Period: Overall Study
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14
Received Treatment | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14
Completed | 5 | 6 | 5 | 6 | 4 | 6 | 6 | 14
Not Completed | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set: all participants who received AMG 570 or the placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.7 (11.4) | 45.8 (14.3) | 43.2 (16.7) | 42.0 (9.8) | 39.8 (17.6) | 39.8 (11.4) | 40.0 (17.1) | 44.4 (12.1) | 43.1 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 9
  Male | 3 | 4 | 5 | 6 | 5 | 6 | 6 | 12 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 4
  Not Hispanic or Latino | 6 | 6 | 5 | 6 | 5 | 6 | 6 | 12 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3 | 0 | 5 | 1 | 3 | 15
  White | 5 | 6 | 3 | 3 | 6 | 1 | 5 | 11 | 40
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced One or More Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were adverse events with an onset after the administration of study treatment.
  TEAEs were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limited age appropriate instrumental activities of daily life (ADL).
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolonged hospitalization indicated; disabling; limited self care ADL.
  Grade 4 Life-threatening consequences; urgent interventions indicated.
  Serious adverse events (SAEs) were defined as meeting at least 1 of the following criteria:
  * Results in death (fatal)
  * Immediately life-threatening
  * Requires in-patient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Other medically important serious event
Time Frame: Day 1 to Day 105
Population: Safety analysis set: all participants who received AMG 570 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14
Participants
  TEAEs | 6 | 5 | 4 | 4 | 2 | 3 | 4 | 9
  Grade ≥ 2 TEAEs | 4 | 0 | 1 | 1 | 0 | 0 | 1 | 3
  Grade ≥ 3 TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade ≥ 4 TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SAEs | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Life-threatening TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatal TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Experienced a Clinically Significant Change in Physical Examinations
Description: Physical examinations were performed by the investigator, designated physician, or nurse practitioner. A complete physical examination included, at a minimum, assessment of cardiovascular, respiratory, gastrointestinal and neurological systems. A brief physical examination included assessment of the skin, lungs, cardiovascular system, and abdomen (liver and spleen).
Time Frame: Baseline to Day 105
Population: Safety analysis set: all participants who received AMG 570 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Who Experienced a Clinically Significant Change in Vital Signs
Description: Any changes in blood pressure, body temperature, heart rate, and pulse rate that were deemed as clinically significant by the Investigator were reported.
Time Frame: Baseline to Day 105
Population: Safety analysis set: all participants who received AMG 570 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Who Experienced a Clinically Significant Change in Clinical Laboratory Safety Tests
Description: Laboratory safety tests included chemistry, hematology, and urinalysis parameters. Clinically significant laboratory safety tests were any events assessed as CTCAE Grade ≥3 at any post-baseline visit.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolonged hospitalization indicated; disabling; limited self care ADL.
  Grade 4 Life-threatening consequences; urgent interventions indicated.
Time Frame: Baseline to Day 105
Population: Safety analysis set: all participants who received AMG 570 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

5. Primary Outcome: Number of Participants Who Experienced a Clinically Significant Change in Electrocardiograms (ECGs)
Description: Any changes in ECG parameters that were deemed clinically significant by the Investigator were reported.
Time Frame: Baseline to Day 105
Population: Safety analysis set: all participants who received AMG 570 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Maximum Observed Concentration (Cmax) of AMG 570
Description: AMG 570 pharmacokinetic (PK) parameters were estimated using non-compartmental analysis.
Time Frame: Pre-dose and 12 hours post-dose on Day 1 and days 2, 3, 4, 6, 8, 11, 15, 22, 29, 43, 57, 71 and 105
Population: The PK concentration analysis set: all participants who received AMG 570 and had at least one quantifiable PK sample collected.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
µg/mL | 0.08664 (0.0539) | 0.624 (0.327) | 4.33 (3.53) | 6.05 (3.26) | 17.2 (3.78) | 33.5 (15.9) | 58.5 (19.9)

7. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of AMG 570
Description: AMG 570 PK parameters were estimated using non-compartmental analysis.
Time Frame: Pre-dose and 12 hours post-dose on Day 1 and days 2, 3, 4, 6, 8, 11, 15, 22, 29, 43, 57, 71 and 105
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
days | 5.0 [2.0 to 5.0] | 3.0 [2.0 to 13] | 3.0 [0.5 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [3.0 to 10] | 5.0 [3.0 to 14] | 5.0 [3.0 to 10]

8. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration (AUClast) of AMG 570
Description: AMG 570 PK parameters were estimated using non-compartmental analysis.
Time Frame: Pre-dose and 12 hours post-dose on Day 1 and days 2, 3, 4, 6, 8, 11, 15, 22, 29, 43, 57, 71 and 105
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: day*µg/mL
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
day*µg/mL | 0.591 (0.321) | 5.12 (2.62) | 43.8 (26.1) | 88.3 (50.1) | 271 (61.3) | 561 (221) | 1660 (759)

9. Secondary Outcome: Area Under the Concentration-time Curve Observed From Time Zero to Infinity (AUCinf) of AMG 570
Time Frame: Pre-dose and 12 hours post-dose on Day 1 and days 2, 3, 4, 6, 8, 11, 15, 22, 29, 43, 57, 71 and 105
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: day*µg/mL
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 5 | 5 | 6
day*µg/mL | 0.928 (0.248) | 6.24 (2.76) | 51.1 (21.9) | 88.6 (50.1) | 284 (59.2) | 624 (176) | 1660 (757)

10. Secondary Outcome: Number of Participants With an Anti-AMG 570 Binding Antibody Positive Postbaseline Result
Description: The presence of anti-AMG 570 binding antibodies was assessed using a validated assay. The number and percentage of participants who developed binding anti-AMG 570 antibodies at any postbaseline visit are presented.
Time Frame: Baseline to Day 105
Population: All participants who received AMG 570 and had a negative or no result for binding antibodies at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 3 | 2 | 1 | 3 | 3 | 6 | 4

11. Secondary Outcome: Mean Peripheral Blood B7-Related Protein-1 (B7RP-1) Receptor Occupancy on Total B Cells
Description: Peripheral B7RP1 (also known as inducible costimulator ligand [ICOSL]) receptor occupancy was calculated from the free ICOSL and total ICOSL measurement from B cells in whole blood.
Time Frame: Day 8; Day 29; Day 57; and Day 105
Population: The pharmacodynamic (PD) analysis set: all participants who had received AMG 570 or placebo and for whom at least one PD parameter had quantifiable baseline sample and a quantifiable PD sample collected at each specified visit.
Measure: Mean (Standard Deviation); unit: Percentage B7RP-1 receptor occupancy
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14
Percentage B7RP-1 receptor occupancy
  Day 8: number analyzed (Participants) | 4 | 5 | 6 | 6 | 6 | 5 | 6 | 14
  Day 8 | 13.73 (8.81) | 43.76 (16.90) | 64.37 (14.80) | 80.82 (6.60) | 88.87 (1.83) | 92.52 (1.52) | 95.97 (1.85) | -0.98 (13.52)
  Day 29: number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 5 | 5 | 14
  Day 29 | 0.36 (19.12) | 20.98 (16.60) | 19.96 (10.94) | 38.30 (9.95) | 72.96 (9.21) | 86.64 (4.12) | 89.60 (9.00) | 0.27 (14.86)
  Day 57: number analyzed (Participants) | 6 | 6 | 5 | 5 | 4 | 5 | 5 | 14
  Day 57 | 3.30 (14.27) | 11.28 (9.20) | 10.14 (8.50) | 6.74 (5.47) | 4.55 (15.36) | 33.20 (20.56) | 65.88 (31.67) | 0.85 (14.42)
  Day 105: number analyzed (Participants) | 5 | 6 | 5 | 6 | 4 | 6 | 6 | 13
  Day 105 | -8.94 (26.16) | 4.53 (10.31) | -4.54 (8.76) | 1.37 (4.45) | -2.25 (8.94) | -0.08 (7.93) | 13.33 (17.05) | -2.90 (15.86)

12. Secondary Outcome: Percentage Change From Baseline for Cluster of Differentiation (CD)19+ Total B Cells Counts
Time Frame: Baseline to Day 8; Day 29; Day 57 and Day 105
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 5 | 6 | 14
Percentage of change
  Percentage change from Baseline at Day 8: number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 5 | 3 | 13
  Percentage change from Baseline at Day 8 | 41.333 (73.517) | 53.770 (43.216) | 66.531 (28.057) | 32.861 (21.296) | 57.123 (75.399) | 57.478 (28.365) | 74.509 (70.354) | 2.671 (20.898)
  Percentage change from Baseline at Day 29: number analyzed (Participants) | 5 | 4 | 5 | 6 | 4 | 5 | 4 | 12
  Percentage change from Baseline at Day 29 | -20.284 (22.310) | -8.084 (10.212) | -17.994 (15.582) | -10.047 (19.791) | 22.735 (51.384) | 26.305 (28.795) | 9.637 (28.555) | 3.031 (23.358)
  Percentage change from Baseline at Day 57: number analyzed (Participants) | 6 | 6 | 5 | 6 | 2 | 5 | 5 | 14
  Percentage change from Baseline at Day 57 | -2.548 (41.873) | -14.215 (14.903) | -27.494 (20.918) | -37.481 (17.440) | 0.386 (50.044) | -8.882 (21.936) | 1.212 (42.870) | 5.726 (28.059)
  Percentage change from Baseline at Day 105: number analyzed (Participants) | 4 | 6 | 3 | 6 | 4 | 5 | 6 | 12
  Percentage change from Baseline at Day 105 | -15.143 (22.117) | 17.010 (33.957) | -16.872 (19.064) | 0.841 (48.458) | -8.111 (32.077) | -24.059 (25.753) | -30.413 (26.863) | 1.023 (13.612)

13. Secondary Outcome: Percentage Change From Baseline for CD19+ Total B Cells Percentages (%)
Time Frame: Baseline to Day 8; Day 29; Day 57 and Day 105
Population: The PD analysis set: all participants who had received AMG 570 or placebo and for whom at least one PD parameters had quantifiable baseline sample and at quantifiable PD sample collected at each specified visit.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 5 | 6 | 14
Percentage of change
  Percentage change from Baseline at Day 8: number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 5 | 3 | 13
  Percentage change from Baseline at Day 8 | 56.111 (88.264) | 24.057 (10.041) | 28.291 (16.950) | 20.942 (7.799) | 26.538 (28.906) | 45.886 (25.595) | 23.693 (21.414) | -1.241 (12.309)
  Percentage change from Baseline at Day 29: number analyzed (Participants) | 5 | 4 | 5 | 6 | 4 | 5 | 4 | 12
  Percentage change from Baseline at Day 29 | -13.714 (17.368) | -13.258 (17.292) | -22.000 (9.603) | -5.778 (12.947) | 2.765 (28.960) | 7.836 (20.250) | 4.063 (15.629) | -0.582 (17.259)
  Percentage change from Baseline at Day 57: number analyzed (Participants) | 6 | 6 | 5 | 6 | 2 | 5 | 5 | 14
  Percentage change from Baseline at Day 57 | 29.484 (84.641) | -21.751 (11.893) | -26.000 (20.346) | -36.293 (18.635) | -16.667 (35.355) | -10.467 (4.058) | -7.500 (19.632) | 0.167 (16.092)
  Percentage change from Baseline at Day 105: number analyzed (Participants) | 4 | 6 | 3 | 6 | 4 | 5 | 6 | 12
  Percentage change from Baseline at Day 105 | -7.738 (8.988) | -1.524 (17.352) | -23.333 (14.530) | -9.947 (17.880) | -15.152 (13.165) | -23.966 (13.136) | -35.474 (10.308) | 3.895 (16.653)

ADVERSE EVENTS:
Time Frame: Up to 105 days
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- AMG 570 - 700 mg: Participants received 700 mg dose of AMG 570 administered as single dose subcutaneous in healthy volunteers.
Arm/Group | AMG 570 - 7 mg | AMG 570 - 21 mg | AMG 570 - 70 mg | AMG 570 - 140 mg | AMG 570 - 210 mg | AMG 570 - 420 mg | AMG 570 - 700 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/14
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 4/6 | 4/6 | 2/6 | 3/6 | 4/6 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 570 - 7 mg (N=6) | AMG 570 - 21 mg (N=6) | AMG 570 - 70 mg (N=6) | AMG 570 - 140 mg (N=6) | AMG 570 - 210 mg (N=6) | AMG 570 - 420 mg (N=6) | AMG 570 - 700 mg (N=6) | Placebo (N=14)
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 570 - 7 mg (N=6) | AMG 570 - 21 mg (N=6) | AMG 570 - 70 mg (N=6) | AMG 570 - 140 mg (N=6) | AMG 570 - 210 mg (N=6) | AMG 570 - 420 mg (N=6) | AMG 570 - 700 mg (N=6) | Placebo (N=14)
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Application site erythema (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Injection site erythema (General disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site warmth (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 2
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT02618967/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT02618967/SAP_001.pdf